CLINICAL TRIAL: NCT00144638
Title: Procalcitonin Increase Identifies Critically Ill Patients at High Risk of Mortality
Status: Completed | Type: Observational
Sponsor: Danish Procalcitonin Study Group (Other)
Other Study IDs: DPSG1
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-02

CONDITIONS: Sepsis - to Reduce Mortality in the Intensive Care Unit

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Procalcitonin, a marker of infection has often been compared to clinical pictures as for instance "clinical sepsis". This has given som problems in the interpretation of these studies, because of the lack of good Gold Standards for "clinical sepsis. We have decided to investigate the development from day to day of Procalcitonin in the blood of intensive care patients, compared to the mortality.

Hypothesis: Procalcitonin increase after reaching a certain level predicts mortality in the Intensive Care Unit.

DETAILED DESCRIPTION:
Sepsis is a major cause of mortality in the Intensive Care Unit (ICU). Efforts have been made to reduce the time needed to diagnose sepsis in order to reduce mortality from sepsis-related multi-organ dysfunction .

Markers of inflammation such as C-reactive protein (CRP) and White Blood Cell count (WBC) have proved far from ideal in identifying critically ill patients who need antimicrobial therapy, because the sensitivity and specificity for bacterial infection is low.

Procalcitonin (PCT) is a 13 kDa 116 amino acid polypeptide, initially described as a prohormone of Calcitonin, a hormone of the calcium metabolism produced in the medullary C-cells of the Thyroid gland5-7. However, recent studies demonstrated that the variant PCT associated with infection can be produced by other tissues.

As kinetic studies on baboons and humans have shown a rapid release within 2-4 hours after injection of bacteria or bacterial toxins, PCT is a substance which is released more rapidly than CRP. The plasma half-life of PCT is close to 24 hours. Measurements of PCT in healthy individuals have shown very low serum levels (<0.05 ng/ml).

In 1993, Assicot et al. reported that elevated levels of serum procalcitonin were closely related to the onset of bacterial infection and seemingly correlated to severity of infection.

Several clinical studies have detected a high PCT level in patients with evidence of systemic bacterial infection, while relatively low PCT levels, on the other hand, occur in patients with only local bacterial infection or viral infection.

Other studies have shown low to only moderately elevated PCT in uninfected patients after major surgery, trauma and after myocardial infarction.

A reduced usage of antimicrobial therapy has been demonstrated when treatment was guided by PCT in patients with suspected lower respiratory tract infection, who were admitted to a medical emergency department. Only few studies, however, have investigated the PCT day-to-day changes for several days in respect of the clinical outcome in a population at risk of contracting serious infections.

The aim of the present study was to assess the ability of PCT-, CRP- and leucocyte measurements in early identification of critically ill patients, who are at high risk of mortality. The study was a one-year study.

Methods Patients From January 2 through December 2002, we conducted an observational study including all patients (except livertransplanted patients) admitted to the multi-disciplinary intensive care unit 4131 at Rigshospitalet, Copenhagen University Hospital, a secondary and tertiary reference hospital. Patients were included on admittance to the ICU. In cases of re-admittance, only measurements from the first admittance were included in the study.

When sepsis was suspected, we performed culture samples from all suspected sites before antibiotic therapy was initiated. Surveillance culture samples were performed twice a week from all patients, including blood cultures from indwelling catheters.

Data of co-morbidity and mortality were registered real-time and were verified via the central hospital register for Rigshospitalet, Copenhagen University Hospital.

In all analyses, mortality was defined as all-cause mortality. The primary endpoint was 90-day survival; secondary endpoints were survival while admitted to the ICU and 30-day survival.

Blood samples Blood samples for PCT measurements were collected by the nursing staff in the ICU on a daily basis between 6.00 a.m. and 7.30 a.m. in accordance with the assumed half life of PCT. PCT analyses were performed by laboratory technicians at the Department of Clinical Microbiology, using an immunoluminometric assay (Lumitest-PCT, B.R.A.H.M.S. Diagnostica, Berlin, Germany). The threshold of detection was 0.1 ng/ml serum, according to the manufacturer.

Blood samples were collected as a routine test in accordance with the ethical procedures of the hospital.

All blood samples were stored at 4o Celsius, and were analysed within maximally 72 hours. As a control of the PCT analysis and storage, we made double determinations. Ten blood samples were analysed single-blinded three times daily at a standardised time for three days.

PCT-day-to-day change analysis Standard empiric antimicrobial treatment of sepsis in this ICU includes: Meropenem and Ciprofloxacin, when relevant supplemented with: Metronidazole, Vancomycin, Linezolid and occasionally other antibiotics according to clinical findings, patient tolerance, suspected site of infection and bacterial cultures from foci and from surveillance cultures combined with susceptibility patterns. Treatment of invasive fungal infection included Caspofungin, Liposomal Amphotericin B or Voriconazole, or combination therapy with these according to Candida species identification and susceptibility pattern from Minimal Inhibitory Concentration (MIC) in surveillance cultures.

ELIGIBILITY:
Inclusion Criteria: Admitted to the ICU 4131 of Rigshospitalet Copenhagen University Hospital in the year 2002

-

Exclusion Criteria:

Recent (< 3 months) liver transplantation

Expected admission < 24 h

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2002-01; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Lars Heslet, MD, MD.Sc., Principal Investigator — Dept. 4131, Rigshospitalet, Blegdamsvej 9, DK-2100
Locations (1):
- Dept. 4131, Rigshospitalet, Cph University Hosp., DK, Copenhagen, Denmark